CLINICAL TRIAL: NCT02741479
Title: The Effectiveness of Kinesio® Tex Tape on Gluteus Medius Activation in Dancers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-00705
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Gluteus Medius Activation
Keywords: dancers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- K Tape Group (Experimental)
  Interventions: Other: Airplane Test
- Sham Group (Active Comparator)
  Interventions: Other: Airplane Test
- No Tape (Experimental)
  Interventions: Other: Airplane Test

INTERVENTIONS:
Other: Airplane Test — The airplane test requires the subject to bend forward, bringing the upper body and one leg horizontal, making a "T" position with the body with the arms out to the sides while in single-leg stance; they then bend the supporting leg, bringing the finger tips towards the floor, followed by straightening the supporting leg and bringing the arms back out to the sides. This motion is repeated five times on each leg per trial. The airplane will be performed to a metronome to standardize performance time

SUMMARY:
The purpose of this research is to determine if a specific type of elasticated athletic tape (Kinesio Tex Tape) increases muscle activation among professional level dancers. Investigators will determine if changes in muscle activation with the elasticated tape differ from changes experienced with no tape and/or sham tape, and if it coincides with subjective sense of muscle activation.

ELIGIBILITY:
Inclusion Criteria:

* Uninjured professional level dancers

Exclusion Criteria:

* Non-professional level of dance or non-dancer; obesity (body mass index greater than 30 kg/m²)
* A history of major back, abdominal, or lower extremity surgery
* A history of muscle diseases; a history of serious cardiovascular diseases (e.g., cardiac insufficiency, arrhythmia, severe hypertension, vascular insufficiency)
* A history of serious respiratory diseases; major fractures of the lower extremities; lower extremity or trunk injury within the last year; a history of surgery within the last year, a history of stroke, acute, or chronic infections; serious metabolic diseases
* Glaucoma
* Structural disease or severe congenital deformities of the spine of a high degree
* Inguinal, femoral, or umbilical hernia; or diseases related to body equilibrium.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Activity measured via electromyography | Baseline and 1.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Donald Rose, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States